CLINICAL TRIAL: NCT05750407
Title: Feasibility of Cardiovascular Health Intervention Within Evidence-based Home Visiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Polytechnic State University-San Luis Obispo (Other)
Collaborators: The Miriam Hospital (Other); Bradley Hospital (Other)
Responsible Party: Principal Investigator, Suzanne Phelan, Professor of Kinesiology & Public Health, California Polytechnic State University-San Luis Obispo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-ENRICH Pilot
Record Dates: First submitted 2023-02-20; First posted 2023-03-01 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Diet, Healthy; Inactivity, Physical; Obesity
Keywords: home visiting; obesity; pregnancy; postpartum; cardiovascular health
MeSH Terms: conditions — Sedentary Behavior; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evidence based home visiting with lifestyle modules (Experimental): Three lifestyle change modules will be discussed with clients: healthy eating, activity, and tracking diet and weight
  Interventions: Behavioral: Lifestyle change

INTERVENTIONS:
Behavioral: Lifestyle change — Three modules target healthy eating, activity, and weight control behaviors

SUMMARY:
The purpose of this pilot study is to examine the feasibility and acceptability of brief lifestyle intervention modules designed to promote healthy eating, activity, and weight control for pregnant and postpartum clients receiving care as part of evidence-based home visiting.

DETAILED DESCRIPTION:
The purpose of this pilot study is to examine the feasibility and acceptability of brief lifestyle intervention modules designed to promote healthy eating, activity, and weight control behaviors for pregnant and postpartum clients receiving care as part of evidence-based home visiting. A 6 week, pre-post test of evidence-based home visiting (usual care) plus three lifestyle intervention modules (eating, activity, tracking) will be conducted at two sites (California and Rhode Island). Three, 10 minute intervention modules will target healthy eating, activity, and self-monitoring of weight and diet. Pregnant and postpartum clients (N =20) in home visiting programs will be recruited over 2 months and evaluated at baseline and after 6 weeks. Home visitors will participate in one training session and deliver the intervention content during three visits over 6 weeks. Quantitative data from will inform feasibility of lifestyle intervention within evidence-based home visiting. Findings will inform the cardiovascular health intervention and study protocol for a full scale trial.

ELIGIBILITY:
Inclusion Criteria:

* self-reported current participation in a home visiting program
* self-reported currently pregnant or postpartum less than or equal to 6 weeks
* English or Spanish speaking

Exclusion Criteria (based on self report):

* Age less than 18 years
* Lower than 5th grade reading level

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Perceived acceptability of treatment score | 6 week
  Questionnaire

SECONDARY OUTCOMES:
Change in life's essential 8 total score | 6 weeks
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cal Poly, San Luis Obispo, California
  - Miriam Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No